CLINICAL TRIAL: NCT04671914
Title: Prevalence of Intrauterine Adhesions After the Application of Hyaluronic Acid Gel After Dilatation and Curettage in Women With Spontaneous Abortion or Induction of Abortion From 12+0 Till 23+6 Week of Pregnancy.
Brief Title: Prevalence of Intrauterine Adhesions After D&C With or Without Antiadhesion Gel After Abortion in Second Trimester.
Acronym: ADAB
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Institute for the Care of Mother and Child, Prague, Czech Republic (Other)
Collaborators: Bulovka Hospital (Other); General University Hospital, Prague (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Intrauterine adhesions 2020
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Asherman Syndrome; Abortion Late
Keywords: Asherman Syndrome; Abortion Late; Hyaluronic acid gel; Hysteroscopy
MeSH Terms: conditions — Gynatresia | interventions — Hyaluronic Acid; Dilatation

STUDY DESIGN:
Intervention Model Description: Multicenter prospective controlled study
Who Masked: Participant, Investigator
Masking Description: Participant will not be informed about usage of hyalobarier gel or not. Care provider - at the time of RCUI the surgeon will know from randomisation if apply the gel or not. The investigator performing evaluation of adhesions by hysteroscopy will be blinded to the arm which the participants belong to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyaluronic acid gel after D&C (Active Comparator): After abortion in the II trimester, we provide D&C and after the procedure, we apply in uterine cavity Hyaluronic acid gel.
  Interventions: Drug: Hyaluronic Acid 20 MG/ML Injectable Solution; Other: Dilation and curretage
- Only D&C (Active Comparator): After abortion, in the II trimester, we provide only D&C.
  Interventions: Other: Dilation and curretage

INTERVENTIONS:
Drug: Hyaluronic Acid 20 MG/ML Injectable Solution — Application of hyaluronic acid gel into uterine cavity after After abortion in II trimester we do D&C
  Arms: Hyaluronic acid gel after D&C
Other: Dilation and curretage — After abortion in II trimester we do D&C.

SUMMARY:
Only patients who sign an informed consent will be included. Patients after a miscarriage in the 2nd trimester of pregnancy who need to perform an instrumental revision of the uterine cavity (RCUI, revisio cavi uteri instrumentalis) will be randomized into two groups. In the first group, RCUI will be performed according to current standards. In the second group, an anti-adhesive preparation with hyaluronic acid (Hyalobarrier gel Endo) will be applied to the uterine cavity at the end of the RCUI procedure. Eight to twelve weeks after the operation, the occurrence of adhesions will be evaluated by ultrasound examination and diagnostic hysteroscopy (if adhesions will be detected, they will be disrupted). The study will also include the completion of a questionnaire in terms of the frequency and strength of the menstrual cycle. The presence of adhesions will be assessed according to The American Fertility Society (AFS).

DETAILED DESCRIPTION:
Methodology Only patients who sign informed consent will be included. Patients after a miscarriage in the 2nd trimester of pregnancy who need to perform an instrumental revision of the uterine cavity (RCUI, revisio cavi uteri instrumentalis) will be randomized into two groups. In the first group, RCUI will be performed according to current standards. In the second group, an anti-adhesive preparation with hyaluronic acid (Hyalobarrier gel Endo) will be applied to the uterine cavity at the end of the RCUI procedure. Eight to twelve weeks after the operation, the occurrence of adhesions will be evaluated by ultrasound examination and diagnostic hysteroscopy (if adhesions will be detected, they will be disrupted). The study will also include the completion of a questionnaire in terms of the frequency and strength of the menstrual cycle. The presence of adhesions will be assessed according to The American Fertility Society (AFS).

Expected number of enrolled subjects: a total of 200 patients, 100 in each branch Entry criteria: Adult (18 to 40 years old) women with a wish for future pregnancy, abortion in the 2nd trimester of pregnancy (over 12 weeks of pregnancy) with instrumental revision of the uterine cavity (RCUI), signed informed consent

Exclusion criteria: age below 18 years, age over 40 years, history of previous uterine surgery (myomectomy, resection of the intrauterine septum, disruption of intrauterine adhesions), suspicion of molar pregnancy, signs of pelvic infection, disagreement with participation in the study

Primary goals of the project:

1. determination of the frequency of intrauterine adhesions in women who underwent instrumental revision of the uterine cavity (RCUI, revisio cavi uteri instrumentalis) after abortion in the 2nd trimester of pregnancy
2. to determine whether the application of an antiadhesive agent with hyaluronic acid has an effect on the frequency of intrauterine adhesions after this procedure

A similar prospective randomized multicenter study investigating the relationship of intrauterine adhesions using an intrauterine gel with hyaluronic acid was published in 2017 by Hooker. Patients were enrolled in the study up to the 14th week of pregnancy. The incidence of intrauterine adhesions was statistically lower in the hyaluronic acid group compared to the no treatment group (13% vs. 30.6%, RR 0.43, 95% CI 0.22-0.83, p 0.013). However, this study investigated RCUI in the first trimester of pregnancy. Our study is to our knowledge the first with a focus on the second trimester RCUI.

Secondary goals of the project:

1. number of pregnancies (pregnancy rate) in the period of 24 months after RCUI in both groups
2. number of term pregnancies in the 24 months after RCUI in both groups

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 to 40 years) women with a wish for future pregnancy
* abortion in the 2nd trimester of pregnancy (over 12 weeks of pregnancy) with instrumental revision of the uterine cavity (RCUI)
* signed informed consent

Exclusion Criteria:

* age below 18 years, age over 40 years
* history of previous uterine surgery (myomectomy, resection of the intrauterine septum, disruption of intrauterine adhesions)
* suspected molar pregnancy
* signs of pelvic infection
* disagreement with participation in the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Intrauterine adhesions after D&C and intrauterine application of hyaluronic acid gell. | 3 month
  To find out wheter the application of antiadhesive agent with hyaluronic acid has an effect on the frequency of intrauterine adhesions after this procedure.
Prevalence of Intrauterine adhesions after D&C. | 3 month
  Dermination of the frequency of intrauterine adhesions in women who underwent instrumental revision of the uterine cavity (RCUI, revisio cavi uteri instrumentalis) after abortion in the 2nd trimester of pregnancy

SECONDARY OUTCOMES:
Pregnancy rate | 24 month
  Number of pregnancies (pregnancy rate) in the period of 24 months after RCUI in both groups
Delivery rate | 24 month
  Number of term deliveries in the 24 months after RCUI in both groups

CONTACTS AND LOCATIONS:
Locations (3):
- Czechia (3):
  - 1.Lf Uk, Vfn, Prague
  - Instiue for Care of Moher and Childe, Prague
  - FN Bulovka, Prague

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang X, Chen C, Wang L, Chen D, Guang W, French J. Conception, early pregnancy loss, and time to clinical pregnancy: a population-based prospective study. Fertil Steril. 2003 Mar;79(3):577-84. doi: 10.1016/s0015-0282(02)04694-0. PMID 12620443
- [Result] Rai R, Regan L. Recurrent miscarriage. Lancet. 2006 Aug 12;368(9535):601-11. doi: 10.1016/S0140-6736(06)69204-0. PMID 16905025
- [Result] ASHERMAN JG. Amenorrhoea traumatica (atretica). J Obstet Gynaecol Br Emp. 1948 Feb;55(1):23-30. doi: 10.1111/j.1471-0528.1948.tb07045.x. No abstract available. PMID 18902559
- [Result] Hooker AB, de Leeuw R, van de Ven PM, Bakkum EA, Thurkow AL, Vogel NEA, van Vliet HAAM, Bongers MY, Emanuel MH, Verdonkschot AEM, Brolmann HAM, Huirne JAF. Prevalence of intrauterine adhesions after the application of hyaluronic acid gel after dilatation and curettage in women with at least one previous curettage: short-term outcomes of a multicenter, prospective randomized controlled trial. Fertil Steril. 2017 May;107(5):1223-1231.e3. doi: 10.1016/j.fertnstert.2017.02.113. Epub 2017 Apr 6. PMID 28390688